CLINICAL TRIAL: NCT03294629
Title: Effects of Pressure Control Device (SensAwake™) on Obstructive Sleep Apnea (OSA) Patients Who Remove the Mask for Unknown Reasons During Automatic Continuous Positive Airway Pressure (Auto-CPAP) Therapy
Brief Title: The Effectiveness of SensAwake™ for Continue Positive Airway Pressure Treatment of Obstructive Sleep Apnea Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 103-7083B
Record Dates: First submitted 2015-08-05; First posted 2017-09-27 (Actual); Results first posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2017-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: cPAP; SenseAwake
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- APAP begins without SensAwake (No Intervention): Patients will receive CPAP treatment without SensAwake™ activation for two weeks, then crossed-over to CPAP treatment with SensAwake™ activation for additional two weeks.
- APAP begins with SensAwake (Experimental): Patients will receive CPAP treatment with SensAwake™ activation for two weeks, then crossed-over to CPAP treatment without SensAwake™ activation for additional two weeks.
  SensAwake™ modification: SensAwake™ is a new design based on the research of Doctor Ayappa 5 years ago. The SensAwake™ modification to the Fisher and Paykel automatically titrating positive airway pressure (APAP) device aims to sense whether the patient is awake via respiratory patterns that differentiate between sleep and wake. Upon sensing that the patient is awake the device is able to reduce positive airway pressure PAP aiming to improve patient comfort which should result in more consolidated sleep.
  Interventions: Device: SensAwake™ modification

INTERVENTIONS:
Device: SensAwake™ modification — SensAwake™ is a new design based on the research of Doctor Ayappa 5 years ago. The SensAwake™ modification to the Fisher and Paykel automatically titrating positive airway pressure (APAP) device aims to sense whether the patient is awake via respiratory patterns that differentiate between sleep and wake. Upon sensing that the patient is awake the device is able to reduce positive airway pressure PAP aiming to improve patient comfort which should result in more consolidated sleep.
  Arms: APAP begins with SensAwake

SUMMARY:
This study will investigate Obstructive Sleep Apnea (OSA) and an automatically Adjusting Positive Airway Pressure (APAP) device with new technology called SensAwake™. This requires experimental confirmation in a randomised controlled trial with crossover design, comparing compliance on standard APAP with compliance using APAP modified by the addition of the SensAwake™ modification on consecutive nights in participants with moderate-to-severe OSA.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be recruited from OSA patients who will remove CPAP himself without any notable reasons.

Exclusion Criteria:

1. Unstable cardiovascular disease (untreated or resistant hypertension acceptable).
2. Inability to tolerate CPAP due to nasal obstruction or claustrophobia as determined by the study investigator.
3. Any known factor or disease that might interfere with treatment compliance, study conduct or interpretation of the results such as psychiatric disease, history of non compliance to medical regimens, or unwillingness to comply with study requirements.
4. Any known factor that result in mask taken of such as skin discomfort, nasal obstruction, water dripping inside the tubing system etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li-Pang Chuang, MD, Principal Investigator — ChangGungMemorialHospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: March 2015 to Mar 2016, at medical clinic.
Groups:
- CPAP w/SensAwake First, Then CPAP w/o SensAwake: Patients will receive CPAP treatment with SensAwake™ activation for two weeks, then crossed-over to CPAP treatment without SensAwake™ activation for additional two weeks. No washout period.
- CPAP w/o SensAwake First, Then CPAP w/SensAwake: Patients will receive CPAP treatment without SensAwake™ activation for two weeks, then crossed-over to CPAP treatment with SensAwake™ activation for additional two weeks. No washout period.
Period: First Intervention (2 Weeks)
Arm/Group | CPAP w/SensAwake First, Then CPAP w/o SensAwake | CPAP w/o SensAwake First, Then CPAP w/SensAwake
Started | 16 | 19
Completed | 14 | 15
Not Completed | 2 | 4
Period: Second Intervention (2 Weeks)
Arm/Group | CPAP w/SensAwake First, Then CPAP w/o SensAwake | CPAP w/o SensAwake First, Then CPAP w/SensAwake
Started | 14 | 15
Completed | 12 | 13
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPAP w/SensAwake First, Then CPAP w/o SensAwake | CPAP w/o SensAwake First, Then CPAP w/SensAwake | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (10.9) | 41.5 (12.0) | 44.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 12 | 10 | 22
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 31.8 (4.3) | 32.9 (6.9) | 32.4 (5.7)
Neck Circumference (NC) [Mean (Standard Deviation); unit: cm] | 42.3 (2.1) | 41.0 (2.2) | 41.6 (2.2)
Apnea-hypopnea index (AHI) [Mean (Standard Deviation); unit: events per hour] — Apnea-hypopnea index is an index used to indicate the severity of sleep apnea. It is represented by the number of apnea and hypopnea events per hour of sleep that recorded in polysomnography.
  events per hour | 55.3 (30.8) | 54.0 (35.3) | 54.6 (32.5)
Sleep efficiency [Mean (Standard Deviation); unit: % (percentage of minutes slept)] — Sleep efficiency is presented by percentage of minutes of sleep divided by the minutes in bed.
  % (percentage of minutes slept) | 82.0 (8.9) | 73.0 (21.3) | 77.1 (17.1)
Total sleep time [Mean (Standard Deviation); unit: minutes] | 301.0 (34.2) | 276.2 (79.2) | 287.6 (62.8)
Deep sleep - Stage 3 [Mean (Standard Deviation); unit: % (percentage of minutes of stage 3)] — Deep sleep is presented by percentage of minutes of stage 3 divided by the minutes of all sleep time.
  % (percentage of minutes of stage 3) | 6.1 (10.4) | 4.4 (5.6) | 5.2 (8.0)
Average used time of CPAP [Mean (Standard Deviation); unit: minutes] | 187.4 (104.6) | 227.9 (104.1) | 208.5 (104.2)
Compliance of CPAP [Mean (Standard Deviation); unit: %] — CPAP compliance is defined as using the therapy for more than 4 hours a night of all the nights.
  % | 31.9 (31.9) | 46.2 (30.6) | 39.3 (31.4)
Residual AHI under CPAP Tx [Mean (Standard Deviation); unit: events per hour] — Apnea-hypopnea index (AHI) is an index used to indicate the severity of sleep apnea. It is represented by the number of apnea and hypopnea events per hour of sleep. Residual AHI is recorded by CPAP device.
  events per hour | 2.9 (1.3) | 4.4 (2.8) | 3.7 (2.3)
Pittsburgh Sleep Quality Index (PSQI) [Mean (Standard Deviation); unit: units on a scale] — The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. Overall score is ranging from 0 to 21, where lower scores denote a healthier sleep quality.
  units on a scale | 7.4 (2.3) | 10.1 (3.8) | 8.8 (3.4)
Epworth Sleepiness Scale (ESS) [Mean (Standard Deviation); unit: units on a scale] — The ESS is a self-administered questionnaire with 8 questions. The ESS score can range from 0 to 24, where higher scores denote a worse daytime sleepiness.
  units on a scale | 13.3 (5.5) | 13.1 (6.7) | 13.2 (6.0)
Nasal Obstruction Symptom Evaluation (NOSE) [Mean (Standard Deviation); unit: units on a scale] — The Nasal Obstruction Symptom Evaluation (NOSE) is a self-administered questionnaire with 11 questions. The NOSE score can range from 0 to 44, where higher scores denote a worse nasal obstruction.
  units on a scale | 13.5 (6.8) | 15.6 (8.4) | 14.6 (7.6)

OUTCOME MEASURES:

1. Primary Outcome: Compliance of Auto-CPAP Therapy
Description: Objective data recorded in the auto-CPAP machine, Percentage of nights of using auto-CPAP for at least 4 hours during therapy.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: percentage of nights
Groups:
- SA ON: CPAP with SensAwake activation
- SA OFF: CPAP without SensAwake activation
Arm/Group | SA ON | SA OFF
Number analyzed (Participants) | 25 | 25
percentage of nights | 41.8 (35.0) | 39.7 (32.6)

2. Secondary Outcome: Average SA Detections
Description: Average detects of arousal per hours. (Objective data recorded in the auto-CPAP machine)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: times/hour
Arm/Group | SA ON | SA OFF
Number analyzed (Participants) | 25 | 25
times/hour | 2.1 (0.9) | 0 (0)

3. Secondary Outcome: Average Pressures of Auto-CPAP Machine
Description: Average Pressures of Auto-CPAP Machine (Objective data recorded in the auto-CPAP machine)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | SA ON | SA OFF
Number analyzed (Participants) | 25 | 25
cmH2O | 6.9 (2.7) | 7.3 (2.6)

4. Secondary Outcome: 90th Percentile Pressures of Auto-CPAP Machine
Description: 90th percentile pressures of auto-CPAP machine (Objective data recorded in the auto-CPAP machine)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | SA ON | SA OFF
Number analyzed (Participants) | 25 | 25
cmH2O | 8.6 (3.0) | 9.2 (2.9)

5. Secondary Outcome: Average Leaks of Auto-CPAP Machine
Description: Average leaks of auto-CPAP machine (Objective data recorded in the auto-CPAP machine)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: liters per minute
Arm/Group | SA ON | SA OFF
Number analyzed (Participants) | 25 | 25
liters per minute | 41.3 (20.1) | 44.6 (22.5)

6. Secondary Outcome: 90th Percentile Leaks of Auto-CPAP Machine
Description: Average leaks of auto-CPAP machine (Objective data recorded in the auto-CPAP machine)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: liters per minute
Arm/Group | SA ON | SA OFF
Number analyzed (Participants) | 25 | 25
liters per minute | 57.6 (24.7) | 58.9 (26.0)

7. Secondary Outcome: Residual Apnea-Hypopnea Index (AHI)
Description: Residual Apnea-Hypopnea index (Objective data recorded in the auto-CPAP machine) means events of apnea and hypopnea per hour during CPAP therapy.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | SA ON | SA OFF
Number analyzed (Participants) | 25 | 25
events per hour | 6.3 (6.7) | 5.0 (4.6)

8. Secondary Outcome: Time Used of Auto-CPAP Machine
Description: Average Time used of auto-CPAP machine (Objective data recorded in the auto-CPAP machine)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | SA ON | SA OFF
Number analyzed (Participants) | 25 | 25
minutes | 213.1 (99.4) | 206.8 (87.6)

9. Secondary Outcome: Percentage of Day Used of Auto-CPAP Machine
Description: Percentage of day used of auto-CPAP machine (Objective data recorded in the auto-CPAP machine)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | SA ON | SA OFF
Number analyzed (Participants) | 25 | 25
Percentage of days | 87.1 (13.8) | 88.1 (11.2)

10. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. Overall score is ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SA ON | SA OFF
Number analyzed (Participants) | 25 | 25
units on a scale | 8.0 (2.6) | 8.0 (2.8)

11. Secondary Outcome: Epworth Sleepiness Score (ESS)
Description: The ESS is a self-administered questionnaire with 8 questions. The ESS score can range from 0 to 24, where higher scores denote a worse daytime sleepiness.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SA ON | SA OFF
Number analyzed (Participants) | 25 | 25
units on a scale | 11.1 (6.1) | 12.1 (7.2)

12. Secondary Outcome: Nasal Obstruction Symptom Evaluation (NOSE)
Description: The Nasal Obstruction Symptom Evaluation (NOSE) is a self-administered questionnaire with 11 questions. The NOSE score can range from 0 to 44, where higher scores denote a worse nasal obstruction.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SA ON | SA OFF
Number analyzed (Participants) | 25 | 25
units on a scale | 14.6 (8.1) | 13.3 (6.7)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | SA ON | SA OFF
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No